CLINICAL TRIAL: NCT05716334
Title: Biosimilars of Rituximab in ANCA-associated Vasculitis Compared to the Originator (BRAVO): a CanVasc Multicentre Study
Brief Title: Biosimilars of Rituximab in ANCA-associated Vasculitis Compared to the Originator
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Sinai Health System (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); St. Joseph's Healthcare Hamilton (Other); University of Calgary (Other); University of British Columbia (Other); University of Alberta (Other); Ottawa Hospital Research Institute (Other); CAnadian Network for Advanced Interdisciplinary Methods for comparative effectiveness research (Unknown); Canadian Initiative for Outcomes in Rheumatology Care (Other)
Responsible Party: Principal Investigator, Arielle Mendel, Assistant Professor, Division of Rheumatology; Clinician Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: MP-37-2021-7545
Record Dates: First submitted 2022-11-30; First posted 2023-02-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: ANCA-associated Vasculitis; Granulomatosis With Polyangiitis; Microscopic Polyangiitis
Keywords: Rituximab; Biosimilar; B-cell depleting therapy; Drug safety; Drug effectiveness
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rituximab originator recipients: Patients aged ≥18 with a diagnosis of GPA or MPA treated with rituximab (RTX) originator for induction and/or maintenance.
- Rituximab biosimilar recipients: Patients aged ≥18 with a diagnosis of GPA or MPA treated with RTX biosimilars (e.g. Ruxience, Truxima, Riximyo, etc) for induction and/or maintenance.

SUMMARY:
The goal of this multicentre observational study is to compare the safety and effectiveness of rituximab biosimilars to the originator in Canadian patients with Granulomatosis with Polyangiitis (GPA) and Microscopic Polyangiitis (MPA), two main forms of ANCA-associated vasculitis (AAV).

The main questions it aims to answer are:

* Is there a difference in vasculitis control between originator and biosimilar rituximab?
* Is there a difference in adverse effects between originator and biosimilar rituximab?
* In the Canadian healthcare context, are wait times to receive approval (financial coverage) for rituximab shorter for biosimilars compared to originators?

Investigators will perform study assessments (including recording disease activity, damage, and adverse events) at the time of participants' usual clinical care visits, at regular intervals for 2 years after starting rituximab (for induction or maintenance treatment) or switching from an originator to a biosimilar as part of their usual care.

Researchers will compare outcomes among participants who have received rituximab originators (from 2018 onwards) or biosimilars as part of their usual care, to see if there are differences in relapses, remission rates, damage, serious infections, serious adverse events, and treatment approval wait times.

DETAILED DESCRIPTION:
Background. Rituximab (RTX), a B-cell depleting therapy, has comparable efficacy to cyclophosphamide for induction of remission in severe granulomatosis with polyangiitis (GPA) and microscopic polyangiitis (MPA) and superior efficacy to azathioprine for maintenance of remission (1,2). RTX is now a first-line therapy for remission induction and maintenance of remission in severe GPA and MPA (3).

Biosimilar RTX agents are molecules that are highly similar in structure to the 'originator' RTX that was initially studied and approved for the treatment of AAV. Among patients with rheumatoid arthritis, randomized controlled trials have demonstrated comparable efficacy and safety between originator and RTX biosimilars (4,5). Extension studies found that switching from originator to biosimilar does not alter disease activity, immunogenicity, or safety (6,7). Conversely, data on the outcomes of RTX biosimilars in AAV are limited. A retrospective study from Korea included 26 patients (~80% MPA) who received either Truxima (n=15) or Mabthera/Rituxan (n=11) for second-line induction after failure or intolerance to cyclosphosphamide (CYC) (8). There were no obvious deviations in relapse, mortality, end-stage kidney disease, or cardiovascular outcomes compared to other studies with similar populations. A second study was a retrospective cohort study of 77 patients with GPA in India who received RTX biosimilars not available in Canada (Reditux, Rituxipca, Mabtas) for induction, maintenance, or both (9). Outcomes were comparable to those observed in randomized controlled trials of the originator drug.

Despite this scarce amount of data, many Canadian provincial and private funders are mandating the use of biosimilar agents (e.g. Truxima, Ruxience, Riximyo) for induction and maintenance of GPA and MPA, in place of the originator drug (Rituxan). There is a need for longitudinal prospective studies to determine comparative safety and effectiveness of RTX biosimilar agents in Canadian patients with GPA or MPA.

The COVID-19 pandemic has raised concerns for patients and providers about the safety of immunosuppression with RTX. Cohort studies of patients with rheumatic disease have reported an association between RTX and the risk of severe COVID-19 and death from COVID-19 (10-12). Rituximab may also reduce the immunogenicity, and thus the effectiveness, of COVID-19 vaccination, as has been observed for other vaccines (13).

Objectives. The overarching objective of this study is to compare the real-world safety and effectiveness of originator and biosimilar RTX for the treatment of GPA/MPA.

Specific objectives:

To determine, in patients with GPA/MPA receiving biosimilar or originator RTX for remission induction and/or maintenance:

1. Frequency of clinical remission at 6 and 24 months
2. Frequency and time to relapse and major relapse at 6 and 24 months
3. Frequency and time to serious adverse events (SAEs) at 6 and 24 months
4. Frequency and time to serious infection (SI) at 6 and 24 months
5. Frequency and time to discontinuation of RTX due to adverse events or relapse
6. Disease damage at 6 and 24 months
7. Wait time from RTX application to approval and first infusion
8. Frequency of COVID-19 infections and hospitalizations

Participant recruitment:

Potential prospective participants meeting inclusion criteria will be identified by clinicians providing care to patients with GPA or MPA (i.e., the local study investigators) when patients attend their routine clinical care visits (in-person or telemedicine). The local study investigators (i.e. the clinician providing care to the patient) will then describe the study to potential participants, and if interested, will be given the informed consent form to read (in paper or electronic format, per the potential participant's wishes). The potential participant will have the opportunity to ask any questions to the clinician/investigator or research coordinator, who will be the person obtaining consent. The potential participant will also have the option of reading the consent form at a later date, and will be given the contact information of the study coordinator should he/she wish to notify the investigator and/or coordinator of his/her intent to participate at a later date.

Informed consent Informed consent will be obtained either electronically (via the secure REDCap platform) or using paper consent forms during usual care visits. Patients' participation is entirely voluntary. Prospective participants will provide informed consent to participate in the study and may discontinue their participation at any time.

This study will be conducted in accord with the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans (2018), as well as in respect of the requirements set out in the applicable standard operation procedures of the Research Institute of the McGill University Health Centre Research Institute and of the McGill University Health Centre Research Ethics Board. The McGill University Health Centre Research Ethics Board has reviewed this study and is responsible for monitoring it at all participating institutions in the health and social services network in Québec. Each participating center outside the Réseau de la Santé et des Services Sociaux has approval from their local Research Ethics Board.

Data Collection

Participants will be followed for 24 months.

The following will be collected at enrolment/baseline:

* Age, sex, race/ethnicity, province, education, diagnosis (GPA or MPA), date of diagnosis, ANCA status at diagnosis, number of prior relapses
* Organ involvement at last relapse or at diagnosis
* Birmingham Vasculitis Activity Score (v3, BVAS) and Vasculitis Damage Index (VDI) at time of RTX treatment
* Prior RTX and cyclophosphamide doses received in the last 5 years, dates
* Type of RTX product received
* Payor (i.e., government drug plan or private insurance or participant out-of-pocket, assessed based on clinical records of drug applications and approvals located in the chart and/or participant report)
* Date of most recent RTX application and date of first infusion
* Current therapies
* Glucocorticoids with current dose
* Other immunosuppressants
* Pneumocystis/infection prophylaxis
* If switching from RTX originator to biosimilar (or vice versa), reason for switch
* COVID-19 infection and vaccination with dates if applicable

Subsequent study assessments Data collection/study visits will occur at Months 3 (+/-1) (RTX induction recipients only) , 6(+/-3), 12(+/-3), and 24(+/-6), coinciding with usual practice clinical care visits.

At these visits, the following information will be recorded, based on physician clinical assessments (participant history, physical exam), and medical chart reviews (outcome definitions are described in Outcomes):

* Interval RTX infusions: doses, dates, RTX product, payor (based on clinical records of drug applications and approvals and/or participant report)
* If RTX infusions were stopped/delayed, reason and date
* Current (ongoing) therapies
* Current GC dose
* Other immunosuppressants
* pneumocystis/infection prophylaxis
* BVAS
* VDI
* Interval disease relapses with date
* Interval serious infections (SIs) with date
* Interval Serious Adverse Events (SAEs) with date
* Symptomatic late onset neutropenia with date
* Symptomatic hypogammaglobulinemia with date
* Interval COVID-19 infection and vaccination with dates
* Date of death and cause of death if applicable

Data will be collected and entered into secure electronic data capture (REDCap) and/or through paper Case Report Forms (for centers without access to REDCap), and subsequently entered centrally in the main study REDCap database.

As this study will be conducted during the COVID-19 pandemic, virtual visits instead of in-person visits will be accepted as they represent the frequent usual care at the time of this pandemic.

Study size rational:

Planned enrollment will be 120 RTX biosimilar users and 120 RTX originator users, either prospectively or from existing registries with retrospective collection, over the course of 18 months, across 8 different participating centres. This study size would provide 80% power (at a significance level of 0.05) to show a 2-fold increase in the percentage with relapses in the biosimilar group, assuming 15% have a relapse at 24 months in the originator group.

Significance Currently very limited data exist on comparative safety or effectiveness of RTX biosimilars versus the originator drug in ANCA-associated vasculitis. This study will provide real-world data on patients receiving either RTX originator or biosimilar for induction or maintenance of GPA or MPA to permit these comparisons.

Funding The study is funded by the Canadian Network for Advanced Interdisciplinary Methods for comparative effectiveness research (CAN-AIM). CAN-AIM has a mandate to compare safety and effectiveness of originator and biosimilar drugs across diseases and disciplines. The study is also funded by the Canadian Initiative for Outcomes in Rheumatology cAre (CIORA), which ultimately aims to improve the care of Canadians diagnosed with a rheumatic disease.

ELIGIBILITY:
Inclusion Criteria:

Prospective cohort:

Initiated within the last 6 months:

1. RTX biosimilar or originator for induction OR
2. RTX biosimilar or originator for maintenance (with or without prior RTX induction) OR
3. Switched from RTX originator maintenance to biosimilar maintenance (4-12 months between infusions)

Historical cohort:

Followed in a prospective longitudinal cohort study/registry within the CanVasc network, and initiated the following after January 1, 2018 but >6 months prior to study enrollment

1. RTX biosimilar or originator for induction OR
2. RTX biosimilar or originator for maintenance (with or without RTX induction)

Exclusion Criteria:

* patients without a diagnosis of GPA or MPA
* patients who did not/are not receiving RTX induction or maintenance therapy
* patients who initiated most recent RTX treatment course prior to Jan 1, 2018
* patients receiving RTX for reasons other than GPA or MPA induction or maintenance (e.g. other concurrent disease)
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 with a diagnosis of GPA or MPA who initiated rituximab (RTX) originator or biosimilar within the last 6 months at the time of enrolment, OR who belong to prospective longitudinal registries and initiated RTX originator or biosimilar after 2018 and > 6 months before enrolment. The limit of January 2018 was chosen to keep the historical cohort as contemporary as possible and limit measurement bias regarding study outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a relapse | 6 months
  Relapse will be defined as active disease in any organ system (BVAS v3>0) after remission had previously been achieved AND need to escalate glucocorticoids (GC) to ≥20 mg/day OR change immunosuppression, including receiving RTX infusion earlier than planned/higher dose than planned
  The proportion of participants with relapses at 6 months will be compared between groups.
Time to relapse | From Month 0 until date of first relapse, assessed up to 24 months
  Relapse will be defined as active disease in any organ system (BVAS v3>0) after remission had previously been achieved AND need to escalate glucocorticoids (GC) to ≥20 mg/day OR change immunosuppression, including receiving RTX infusion earlier than planned/higher dose than planned.
  Survival analyses will compare time to disease relapse between originator and biosimilar recipients, adjusting for potential confounders

SECONDARY OUTCOMES:
Proportion of participants with a major relapse | 6 months
  Major relapse will be defined as any relapse with one or more of the BVAS/WG major items: gangrene, scleritis, retinal exudates/hemorrhage, sensorineural deafness, mesenteric ischemia, alveolar hemorrhage, respiratory failure, urinary red blood cell casts, rise in creatinine >30% or fall in creatinine clearance >25%, meningitis, cord lesion, stroke, cranial nerve palsy, sensory peripheral neuropathy, motor mononeuritis multiplex
  The proportion of participants with a major relapse at 6 months will be compared between groups.
Proportion in clinical remission 6 months post-induction | 6 months
  Assessed in subgroup receiving RTX induction. Clinical remission will be defined as absence of disease activity in any organ system (BVAS v3=0)
Proportion with a Serious Adverse Event (SAE) | 6 months
  SAE will be defined as any medical event, not necessarily causally related to the treatment, that requires inpatient hospitalization, prolongation of hospitalization, causes a congenital malformation, results in significant disability or incapacity, that is life threatening or that results in death. Sensitivity analysis will exclude hospitalizations due to disease relapse as SAEs.
  The proportion of participants with >=1 SAE will be compared between groups at 6 months.
Proportion with a Serious Infection (SI) | 6 months
  SI will be defined as any infection requiring intravenous (IV) antibiotics, or resulting in hospitalization, prolonging hospitalization, or death
  The proportion of participants with >=1 SI will be compared between groups at 6 months. Survival analyses will compare time to SI between biosimilar and originator groups, adjusting potential confounders and stratifying by RTX exposure type (induction only vs induction + maintenance).
Wait time (days) from RTX application to approval and first infusion | 6 months
  Among participants newly starting RTX for induction or maintenance, mean wait time from RTX application to approval and infusion will be compared between originator and biosimilar groups using multiple linear regression, adjusting for potential confounders.
  Secondary analyses will stratify outcomes according RTX exposure category (RTX induction only, RTX induction followed by RTX maintenance, RTX maintenance without RTX induction).
Change in Vasculitis Damage Index (VDI) | From Baseline (Month 0) to 6 months
  Vasculitis damage will be measured with the Vasculitis Damage Index (VDI).
  Change in VDI over time will be compared between groups using linear mixed effects models for repeated measures, overall and according RTX exposure category (RTX induction only, RTX induction followed by RTX maintenance, RTX maintenance without RTX induction).
Proportion with a Relapse | 24 months
  Relapse will be defined as active disease in any organ system (BVAS v3>0) after remission had previously been achieved AND need to escalate glucocorticoids (GC) to ≥20 mg/day OR change immunosuppression, including receiving RTX infusion earlier than planned/higher dose than planned.
  The proportion of participants with >=1 relapse at 24 months will be compared between originator and biosimilar recipients.
Proportion with Major relapse | 24 months
  Major relapse will be defined as any relapse with one or more of the BVAS/WG major items: gangrene, scleritis, retinal exudates/hemorrhage, sensorineural deafness, mesenteric ischemia, alveolar hemorrhage, respiratory failure, urinary red blood cell casts, rise in creatinine >30% or fall in creatinine clearance >25%, meningitis, cord lesion, stroke, cranial nerve palsy, sensory peripheral neuropathy, motor mononeuritis multiplex
  The proportion of participants with >=1 major relapse at 24 months will be compared between originator and biosimilar groups.
Proportion with a Serious Adverse Event (SAE) | 24 months
  SAE will be defined as any medical event, not necessarily causally related to the treatment, that requires inpatient hospitalization, prolongation of hospitalization, causes a congenital malformation, results in significant disability or incapacity, that is life threatening or that results in death. Sensitivity analysis will exclude hospitalizations due to disease relapse as SAEs.
  The proportion of participants with >=1 SAE will be compared between groups at 24 months.
Proportion with a Serious Infection (SI) | 24 months
  SI will be defined as any infection requiring intravenous (IV) antibiotics, or resulting in hospitalization, prolonging hospitalization, or death
  The proportion of participants with >=1 SI will be compared between groups at 24 months.
Proportion needing to discontinue RTX due to treatment failure | 24 months
  Treatment failure is defined as rituximab cessation due to an adverse event or relapse. The proportion discontinuing RTX due to treatment failure (due to adverse events or relapse) will be compared between groups.
Change in Vasculitis Damage Index (VDI) | From Baseline (Month 0) to 24 months
  Vasculitis damage will be measured with the Vasculitis Damage Index (VDI).
  Change in VDI over time will be compared between groups using linear mixed effects models for repeated measures, overall and according RTX exposure category (RTX induction only, RTX induction followed by RTX maintenance, RTX maintenance without RTX induction).
Time to major relapse | From Month 0 until date of first major relapse, assessed up to 24 months
  Major relapse will be defined as any relapse with one or more of the BVAS/WG major items: gangrene, scleritis, retinal exudates/hemorrhage, sensorineural deafness, mesenteric ischemia, alveolar hemorrhage, respiratory failure, urinary red blood cell casts, rise in creatinine >30% or fall in creatinine clearance >25%, meningitis, cord lesion, stroke, cranial nerve palsy, sensory peripheral neuropathy, motor mononeuritis multiplex
  Survival analyses will compare time to major relapse between originator and biosimilar recipients.
Time to Serious Adverse Event (SAE) | From baseline (Month 0) until date of first SAE, assessed up to 24 months
  SAE will be defined as any medical event, not necessarily causally related to the treatment, that requires inpatient hospitalization, prolongation of hospitalization, causes a congenital malformation, results in significant disability or incapacity, that is life threatening or that results in death. Sensitivity analysis will exclude hospitalizations due to disease relapse as SAEs.
  Survival analyses will compare time to SAE between exposure groups, adjusting for potential confounders
Time to Serious Infection (SI) | From baseline (Month 0) until date of first SI, assessed up to 24 months
  SI will be defined as any infection requiring intravenous (IV) antibiotics, or resulting in hospitalization, prolonging hospitalization, or death
  Survival analyses will compare time to SI between biosimilar and originator groups, adjusting potential confounders and stratifying by RTX exposure type (induction only vs induction + maintenance).
Time to RTX discontinuation due to treatment failure | From Month 0 until date of first relapse, assessed up to 24 months
  Treatment failure is defined as rituximab cessation due to an adverse event or relapse.
  Survival analyses will compare time to RTX discontinuation due to adverse event or relapse between originator and biosimilar groups.

OTHER OUTCOMES:
COVID-19 infections | 6 months
  Rates of COVID-19 infections will be assessed among participants treated with RTX from September 2019 onwards (either originator or biosimilar, induction or maintenance), overall and stratified by vaccination status
COVID-19 hospitalizations | 6 months
  Rates of COVID-19 hospitalizations at 6 months will be assessed among participants treated with RTX from September 2019 onwards (either originator or biosimilar, induction or maintenance), overall and stratified by vaccination status
COVID-19 infections | 24 months
  Rates of COVID-19 infections will be assessed among participants treated with RTX from September 2019 onwards (either originator or biosimilar, induction or maintenance), overall and stratified by vaccination status
COVID-19 hospitalizations | 24 months
  Rates of COVID-19 hospitalizations at 24 months will be assessed among participants treated with RTX from September 2019 onwards (either originator or biosimilar, induction or maintenance), overall and stratified by vaccination status
Symptomatic late onset neutropenia (LON) | 24 months
  Symptomatic late onset neutropenia (LON) is defined as neutropenia associated with fever OR infection where no other explanation is found (LON typically occurs a month after the RTX infusion, and is most often totally asymptomatic).
  Crude event rates of LON will be calculated by dividing the number of events during follow-up by the corresponding person-time at risk.
Symptomatic hypogammaglobulinemia | 24 months
  Symptomatic hypogammaglobulinemia is defined as infection associated with hypogammaglobulinemia (IgG < local laboratory limit).
  Crude event rates of symptomatic hypogammaglobulinemia in each exposure group will be calculated by dividing the number of events during follow-up by the corresponding person-time at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Mendel, MD MSc, Principal Investigator — McGill University
Locations (9):
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia (Vancouver Coastal Health Authority), Vancouver, British Columbia
  - St Joseph's Healthcare Hamilton (McMaster University), Hamilton, Ontario
  - Lawson Research Institute (Western University), London, Ontario
  - Ottawa Hospital Research Institute (Ottawa University), Ottawa, Ontario
  - Sinai Health System (University of Toronto), Toronto, Ontario
  - McGill University (Montreal General Hospital), Montreal, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux du Nord-de-l'île-de-Montréal (CIUSSS NÎM) / Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Guillevin L, Pagnoux C, Karras A, Khouatra C, Aumaitre O, Cohen P, Maurier F, Decaux O, Ninet J, Gobert P, Quemeneur T, Blanchard-Delaunay C, Godmer P, Puechal X, Carron PL, Hatron PY, Limal N, Hamidou M, Ducret M, Daugas E, Papo T, Bonnotte B, Mahr A, Ravaud P, Mouthon L; French Vasculitis Study Group. Rituximab versus azathioprine for maintenance in ANCA-associated vasculitis. N Engl J Med. 2014 Nov 6;371(19):1771-80. doi: 10.1056/NEJMoa1404231. PMID 25372085
- [Background] Mendel A, Ennis D, Go E, Bakowsky V, Baldwin C, Benseler SM, Cabral DA, Carette S, Clements-Baker M, Clifford AH, Cohen Tervaert JW, Cox G, Dehghan N, Dipchand C, Dhindsa N, Famorca L, Fifi-Mah A, Garner S, Girard LP, Lessard C, Liang P, Noone D, Makhzoum JP, Milman N, Pineau CA, Reich HN, Rheaume M, Robinson DB, Rumsey DG, Towheed TE, Trudeau J, Twilt M, Yacyshyn E, Yeung RSM, Barra LB, Khalidi N, Pagnoux C. CanVasc Consensus Recommendations for the Management of Antineutrophil Cytoplasm Antibody-associated Vasculitis: 2020 Update. J Rheumatol. 2021 Apr;48(4):555-566. doi: 10.3899/jrheum.200721. Epub 2020 Sep 15. PMID 32934123
- [Background] Smolen JS, Cohen SB, Tony HP, Scheinberg M, Kivitz A, Balanescu A, Gomez-Reino J, Cen L, Zhu P, Shisha T. A randomised, double-blind trial to demonstrate bioequivalence of GP2013 and reference rituximab combined with methotrexate in patients with active rheumatoid arthritis. Ann Rheum Dis. 2017 Sep;76(9):1598-1602. doi: 10.1136/annrheumdis-2017-211281. Epub 2017 Jun 21. PMID 28637670
- [Background] Park W, Bozic-Majstorovic L, Milakovic D, Berrocal Kasay A, El-Khouri EC, Irazoque-Palazuelos F, Molina FFC, Shesternya P, Miranda P, Medina-Rodriguez FG, Wiland P, Jeka S, Chavez-Corrales J, Garmish O, Linde T, Rekalov D, Hrycaj P, Krause A, Fomina N, Piura O, Abello-Banfi M, Suh CH, Shim SC, Lee SJ, Lee SY, Kim SH, Yoo DH. Comparison of biosimilar CT-P10 and innovator rituximab in patients with rheumatoid arthritis: a randomized controlled Phase 3 trial. MAbs. 2018 Aug/Sep;10(6):934-943. doi: 10.1080/19420862.2018.1487912. Epub 2018 Jul 16. PMID 30010481
- [Background] Cohen SB, Burgos-Vargas R, Emery P, Jin B, Cronenberger C, Vazquez-Abad MD. Extension Study of PF-05280586, a Potential Rituximab Biosimilar, Versus Rituximab in Subjects With Active Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2018 Nov;70(11):1598-1606. doi: 10.1002/acr.23586. PMID 29692005
- [Background] Park W, Suh CH, Shim SC, Molina FFC, Jeka S, Medina-Rodriguez FG, Hrycaj P, Wiland P, Lee EY, Shesternya P, Kovalenko V, Myasoutova L, Stanislav M, Radominski S, Lim MJ, Choe JY, Lee SJ, Lee SY, Kim SH, Yoo DH. Efficacy and Safety of Switching from Innovator Rituximab to Biosimilar CT-P10 Compared with Continued Treatment with CT-P10: Results of a 56-Week Open-Label Study in Patients with Rheumatoid Arthritis. BioDrugs. 2017 Aug;31(4):369-377. doi: 10.1007/s40259-017-0233-6. PMID 28600696
- [Background] Kwon HC, Kim MK, Song JJ, Park YB, Lee SW. Rituximab Biosimilar Prevents Poor Outcomes of Microscopic Polyangiitis and Granulomatosis with Polyangiitis as Effectively as Rituximab Originator. Yonsei Med J. 2020 Aug;61(8):712-719. doi: 10.3349/ymj.2020.61.8.712. PMID 32734735
- [Background] Mittal S, Naidu GSRSNK, Jha S, Rathi M, Nada R, Minz RW, Sharma K, Dhir V, Jain S, Sharma A. Experience with similar biologic rituximab in 77 patients of granulomatosis with polyangiitis-a real-life experience. Clin Rheumatol. 2021 Feb;40(2):645-651. doi: 10.1007/s10067-020-05261-7. Epub 2020 Jul 12. PMID 32656662
- [Background] Loarce-Martos J, Garcia-Fernandez A, Lopez-Gutierrez F, Garcia-Garcia V, Calvo-Sanz L, Del Bosque-Granero I, Teran-Tinedo MA, Boteanu A, Bachiller-Corral J, Vazquez-Diaz M. High rates of severe disease and death due to SARS-CoV-2 infection in rheumatic disease patients treated with rituximab: a descriptive study. Rheumatol Int. 2020 Dec;40(12):2015-2021. doi: 10.1007/s00296-020-04699-x. Epub 2020 Sep 18. PMID 32945944
- [Background] FAI2R /SFR/SNFMI/SOFREMIP/CRI/IMIDIATE consortium and contributors. Severity of COVID-19 and survival in patients with rheumatic and inflammatory diseases: data from the French RMD COVID-19 cohort of 694 patients. Ann Rheum Dis. 2021 Apr;80(4):527-538. doi: 10.1136/annrheumdis-2020-218310. Epub 2020 Dec 2. PMID 33268442
- [Background] Strangfeld A, Schafer M, Gianfrancesco MA, Lawson-Tovey S, Liew JW, Ljung L, Mateus EF, Richez C, Santos MJ, Schmajuk G, Scire CA, Sirotich E, Sparks JA, Sufka P, Thomas T, Trupin L, Wallace ZS, Al-Adely S, Bachiller-Corral J, Bhana S, Cacoub P, Carmona L, Costello R, Costello W, Gossec L, Grainger R, Hachulla E, Hasseli R, Hausmann JS, Hyrich KL, Izadi Z, Jacobsohn L, Katz P, Kearsley-Fleet L, Robinson PC, Yazdany J, Machado PM; COVID-19 Global Rheumatology Alliance. Factors associated with COVID-19-related death in people with rheumatic diseases: results from the COVID-19 Global Rheumatology Alliance physician-reported registry. Ann Rheum Dis. 2021 Jul;80(7):930-942. doi: 10.1136/annrheumdis-2020-219498. Epub 2021 Jan 27. PMID 33504483
- [Background] Rondaan C, Furer V, Heijstek MW, Agmon-Levin N, Bijl M, Breedveld FC, D'Amelio R, Dougados M, Kapetanovic MC, van Laar JM, Ladefoged de Thurah A, Landewe R, Molto A, Muller-Ladner U, Schreiber K, Smolar L, Walker J, Warnatz K, Wulffraat NM, van Assen S, Elkayam O. Efficacy, immunogenicity and safety of vaccination in adult patients with autoimmune inflammatory rheumatic diseases: a systematic literature review for the 2019 update of EULAR recommendations. RMD Open. 2019 Sep 9;5(2):e001035. doi: 10.1136/rmdopen-2019-001035. eCollection 2019. PMID 31565247